CLINICAL TRIAL: NCT06947967
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Multicenter Study of Tucidinostat in Combination With CHOP in Newly Diagnosed Peripheral T-Cell Lymphoma With Follicular Helper of T Cell Phenotype (SWIFT 02)
Brief Title: Tucidinostat in Combination With CHOP in Newly Diagnosed Peripheral T-Cell Lymphoma With Follicular Helper of T Cell Phenotype
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDM304
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-CHOP (Experimental)
  Interventions: Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone); Drug: Tucidinostat
- CHOP (Placebo Comparator)
  Interventions: Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone); Drug: Placebo

INTERVENTIONS:
Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone) — Cyclophosphamide 750 mg/m2 , intravenous infusion on day 1 of each 21-day cycle. Doxorubicin 70mg/m2 , intravenous infusion on day 1 of each 21-day cycle, total 6 cycles. Vincristine 1.4mg/m2(Max dose 2mg), intravenous injection on day 1 of each 21-day cycle , total 6 cycles. Prednisone 100 mg, oral, day 1-5 of each 21-day cycle,total 6 cycles.
Drug: Tucidinostat — oral, taking as prescribed by the protocol
  Arms: C-CHOP
Drug: Placebo — oral, taking as prescribed by the protocol
  Arms: CHOP

SUMMARY:
A Randomised, Double-blind, Multicenter Phase Ⅲ Study to Evaluate the Efficacy and Safety of Tucidinostat versus Placebo in Combination with CHOP in Newly Diagnosed Peripheral T-Cell Lymphoma with Follicular Helper of T Cell Phenotype

DETAILED DESCRIPTION:
This is A Randomised, Double-blind, Multicenter Phase Ⅲ Study to Evaluate the Efficacy and Safety of Tucidinostat versus Placebo in Combination with CHOP in Newly Diagnosed Peripheral T-Cell Lymphoma with Follicular Helper of T Cell Phenotype.Participants Will be Randomised (1:1) to ReceiveTucidinostat (Experimental Arm) or Placebo(Control Arm)in Combination with CHOP .

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent for the study.
2. Male or female, age ≥ 18 years and ≤80 years.
3. ECOG PS 0,1 or 2.
4. Participants with histologically proven peripheral T-cell lymphoma with T-follicular helper phenotype (PTCL-TFH), including: a. angioimmunoblastic T-cell lymphoma, b. follicular helper T-cell lymphoma, follicular type, c. follicular helper T-cell lymphoma, NOS.
5. At least one measurable disease according to the Lugano 2014 Classification.
6. Laboratory criteria are as follows except that caused by lymphoma assessed by the investigator (without receiving any supportive treatment for the following parameters within 2 weeks from the last dose prior to study entry):

(1)Hematology values:Hemoglobin (Hb)≥90g/L,Absolute neutrophil count (ANC) ≥1.5×10 9/L, platelets ≥90×10 9/L (2)Biochemical values: Serum creatinine ≤1.5×upper limit of normal(ULN),Total bilirubin ≤1.5 × ULN, Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) ≤2.5×ULN(ALT, AST≦5×ULN if liver involved).

7.Expected survival≥6 months.

Exclusion Criteria:

1. Presence of CNS involvement.
2. Received prior therapies targeting lymphoma.
3. Participants planned for autologous or allogeneic transplant as consolidation after CR.
4. Participants with any other malignancy in past 5 years, except for local tumors that have been cured.
5. Prior treatment with cytotoxic drugs for another condition (e.g., rheumatoid arthritis).
6. Any investigational therapy within 3 months.
7. Contraindication to any of the individual components of CHOP.
8. Corticosteroid use > 30 mg/day of prednisone or equivalent, for purposes other than lymphoma symptom control, and the following conditions for inclusion must be met, a. participants receiving corticosteroid treatment with ≤ 30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to randomization, b. If glucocorticoid treatment is urgently required for lymphoma symptom control prior to the start of study treatment, prednisone 100 mg or equivalent could be given for a maximum of 7 days, but all tumor assessments must be completed prior to start of glucocorticoid treatment.
9. Ongoing serious central nervous system disease or peripheral neuropathy, such as progressive multifocal leukoencephalopathy.
10. Have uncontrolled or significant cardiovascular disease, including a. Grade Ⅱ or higher Congestive heart failure, unstable angina pectoris, myocardial infarction (New York Heart Association Functional Classification ) within 6 months prior to study entry; or arrhythmia requiring treatment, or Left Ventricular Ejection Fraction (LVEF) < 50% during screening stage b.Primary cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al) c.History of significant QT interval prolongation, or Corrected QT Interval QTc≥450ms(male), QTc≥470ms（female）at screening d.Symptomatic coronary heart disease requiring treatment e.Any other cardiovascular disease which is inappropriate for the study according to investigators' judgment.
11. History of interstitial lung disease(ILD), or with ongoing signs and symptoms by CT or MRI at the time of screening.
12. Participants with factors that could affect oral medication (such as dysphagia, chronic diarrhea, intestinal obstruction etc), or undergone gastrectomy.
13. History of deep vein thrombosis or pulmonary embolism.
14. History of active bleeding within 2 months prior to the start of Cycle 1;or participants receiving anticoagulation therapy; or participants with evidence of bleeding potential according to investigators' judgment ( esophageal varices, active ulcer, or fecal occult blood test positive etc. ). participants with bleeding led by lymphoma according to investigators' judgment are eligible.
15. Major surgical procedures (craniotomy, thoracotomy, or laparotomy) or severe unhealed wounds, ulcers, or fractures were performed within 4 weeks. Tissue biopsy or other minor surgical procedure (other than venipuncture for intravenous fluids) within 7 days.
16. Active infection requiring systemic treatment (oral, intravenous infusion) was present within 2 weeks prior to the first dose. Participants receiving prophylactic antibiotic therapy (e.g., interstitial pneumonia) may be enrolled.
17. HBsAg or HBcAb positive with virus replication (except for virus replication positive that non-active hepatitis B assessed by investigators), HCV-Ab positive with virus replication positive, active syphilis infection (positive for syphilitic-specific and non-specific antibodies).
18. History of HIV infection, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation or stem cell transplantation.
19. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document, or limit compliance with study requirements/ treatment.
20. Drug or alcohol abuse.
21. Women patients of childbearing potential who are unwilling or unable to use an effective method of contraception throughout the treatment period of this trial and for 12 weeks after the last dose of tucidinostat/placebo or CHOP, whichever is the latest, or the spouses of male participants.
22. Any other condition which is inappropriate for the study according to investigators' judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 60 month
  Defined as the duration from the date of randomization to the date of progression, relapse from CR, or death, whichever occurred first.

SECONDARY OUTCOMES:
Complete Response Rate(CRR) | Up to approximately 36 months
Overall response rate (ORR) | Up to approximately 36months
  Defined as the proportion of subjects with measurable disease who achieve CR or partial response (PR)
Event Free Survival (EFS) | Up to approximately 60 month
  Defined as the duration from the date of randomization to the date of disease progression, initiation of subsequent systemic antilymphoma therapy for residual disease, or death, whichever occurs first.
Disease-Free Survival (DFS) | Up to approximately 60 month
  Defined for participants achieving CR as the period from the date of the initial CR until the date of relapse or death from any cause.
Overall Survival (OS) | Up to approximately 60 month
  defined as the duration from the date of randomization to the date of the participant's death
Safety and Tolerability | Up to approximately 78 months
  Number of Participants Who Experience an Adverse Event (AE) assessed by CTCAE v5.0.
Plasma concentrations of tucidinostat | Up to approximately 60 month
  Plasma samples were collected from the participants at the defined time points. Plasma concentrations were measured using a validated, specific, and sensitive method.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No